CLINICAL TRIAL: NCT00004727
Title: African American Antiplatelet Stroke Prevention Study
Brief Title: Antiplatelet Therapy to Prevent Stroke in African Americans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: R01NS033430 (NIH)
Record Dates: First submitted 2000-02-25; First posted 2000-02-28 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Stroke; Cerebral Infarction
Keywords: African American; antiplatelet; aspirin; ASA; acetylsalicylic acid; ticlopidine; prevention; stroke; cerebral infarction; Chicago; non-cardioembolic ischemic stroke
MeSH Terms: conditions — Stroke; Cerebral Infarction | interventions — Aspirin; Ticlopidine

INTERVENTIONS:
Drug: aspirin
Drug: ticlopidine

SUMMARY:
The African-American Antiplatelet Stroke Prevention Study is designed to prevent recurrent strokes by administration of aspirin or ticlopidine. The study also provides community information on reducing risk of stroke and recognizing the symptoms of stroke. The study involves more than 50 participating hospitals located throughout the United States. Study medication is provided free of charge, and a transportation stipend is available for those in need.

DETAILED DESCRIPTION:
Stroke is one of the important diseases that disproportionately affects African-Americans. African-American men and women are about 2 times more likely than whites to die of cerebrovascular disease or experience stroke. Scientific information about the efficacy and safety of stroke preventatives in this group is much needed, yet African-Americans and other minorities have been underrepresented in biomedical research studies. Preliminary data collected from nonwhite, predominantly African-American patients, suggest that ticlopidine is more effective than aspirin in the secondary prevention of stroke and death for these patients and that the risk of serious adverse events is lower. This is a multicenter, randomized, double-blind clinical trial of ticlopidine hydrochloride (500mg/day) and aspirin (650mg/day) in African-American patients with recent non-cardioembolic ischemic stroke. The primary purpose of the study is to compare the efficacy of ticlopidine and aspirin in the prevention of the outcome endpoints recurrent stroke, vascular death, and myocardial infarction in these African-American patients. Adverse experiences will be studied to further our understanding of the safety of these medications in this group. The study is being conducted at 50 sites experienced in the diagnosis and treatment of stroke. 1800 patients are being enrolled over 3-5 years, and each will be in the study for at least 2 years. Patients will be randomly assigned to treatment at least 7 days, but no more than 90 days after cerebral infarction. The trial promises to provide much needed information about secondary stroke prevention in African-Americans and has the support of established African-American physician, church-based, and community organizations. Enrollment of a substantial number of African-American women is anticipated. Data from these patients will significantly add to our understanding of cerebrovascular disease among black women. Furthermore, the study could also serve as an organizational framework for future studies of stroke prevention or hyperacute treatment in the African-American population.

ELIGIBILITY:
Inclusion Criteria:

* African Americans are eligible if they had a non-cardioembolic ischemic stroke at lease 7 days, but no more than 90 days before entering the trial.
* African American
* 29-85 years of age
* Non-cardioembolic cerebral infarct
* Onset of entry stroke at least 7 days but no more than 90 days
* CT or MRI following entry stroke and consistent with occurrence of entry stroke (i.e., shows entry infarct, shows old infarct, or shows no infarct) Measurable neurologic deficit that correlates with onset of entry stroke.
* Informed consent
* Able to follow outpatient treatment program

Exclusion Criteria:

* Volunteers with transient ischemic attack (TIA) as the potentially qualifying event, intracranial hemorrhage, nonatherosclerotic stroke, sensitivity or major allergy to the study drugs, Modified Barthel Index < 10 or childbearing potential are not eligible.
* Non-qualifying entry events: TIA, subarachnoid hemorrhage, cardiac embolism, iatrogenic stroke, postoperative stroke within 30 days of operation, and carotid endarterectomy as preventive treatment of entry stroke.
* Mean arterial blood pressure > 130mmHg on 3 consecutive days
* Modified Barthel Index < 10
* History of dementia or neurodegenerative disease
* Severe comorbid condition such as cancer that would limit survival during 2 year follow-up period
* Concurrent enrollment in another clinical trial
* Sensitivity or allergy to aspirin or ticlopidine
* Women of childbearing potential
* Peptic ulcer disease, active bleeding diathesis, lower gastrointestinal bleeding, platelet or other hematologic abnormality currently active or clinically active in the past year, hematuria, positive stool guaiac, prolonged PT or PTT, BUN > 40mg%, serum creatinine > 2.0mg%, thrombocytopenia or neutropenia as defined by the lower limit of normal for the platelet count or white blood cell count, respectively (absolute neutrophil count of > 1800/mm3 required for participation), or > 2 times the upper range of normal on liver function tests (SGOT, SGPT, total bilirubin)

Ages: 29 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Philip B. Gorelick, M.D., M.P.H, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois, United States